CLINICAL TRIAL: NCT07365878
Title: Effect of Dry Needling on Insulin Resistance in Obese Post- Menopausal Women
Brief Title: Effect of Dry Needling on Insulin Resistance in Obese Post Menopausal Women
Acronym: Dry needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Mohammed Abdo Mohammed, principle investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006055
Record Dates: First submitted 2025-12-14; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance-abdominal Fats -Post Menopausal Women

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needle (Experimental): 26 patients who were treated with Dry Needling (three times /week/4 months), abdominal exercises, and medical standard care for insulin resistance.
  Interventions: Other: Dry Needle; Other: abdominal exercises, and medical standard care for insulin resistance
- abdominal exercises and medical standard care for insulin resistance. (Other): While Group (B), 26 patients treated with abdominal exercises and medical standard care for insulin resistance.
  Interventions: Other: abdominal exercises, and medical standard care for insulin resistance

INTERVENTIONS:
Other: Dry Needle — Dry Needle has been used to treat obesity. Clinical research has found that it is particularly effective for abdominal fat loss.Dry needling in the abdominal region requires an in-depth understanding of the underlying anatomy due to significant safety risks.
  Arms: Dry Needle
Other: abdominal exercises, and medical standard care for insulin resistance — To reduce belly fat, combine core-strengthening exercises like planks, bicycle crunches, and leg raises with overall fat-burning cardio (walking, running) and a healthy diet

SUMMARY:
The aim of the study is to determine the effect Dry Needling of on insulin resistance in obese postmenopausal women.

DETAILED DESCRIPTION:
Insulin resistance and abdominal obesity have a negative impact on quality of life of postmenopausal women. Obesity and, more specifically, the level of intra-abdominal fat, are positively associated with cardiovascular disease and cardiovascular disease risk factors such as increased plasma lipids and lipoproteins, hyperinsulinemia, and insulin resistance. This study has shown associations among menopause, body fat, and body fat distribution, suggesting that increased abdominal fat distribution could partially mediate the increased cardiovascular disease risk of postmenopausal women .

Abdominal obesity can reflect excess of visceral fat tissue or subcutaneous or both. Visceral fat contributes to the pathogenesis of glucose intolerance and insulin resistance. Insulin resistance is an impaired condition of glucose absorption that induced by insulin .It represents a significant medical and socioeconomic issue impacting women's health and quality of life. So there is clinical experience and documentation for the effectiveness of Dry Needling in the treatment of insulin resistance in obese post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* • All participants post-menopausal from at least 3 years.

  * All participants' ages will be ranged from 48-60 years old.
  * All participants BMI will exceed 25-30 kg/m2.
  * All participants waist hip ratio will be equal or more than 0, 90.

Exclusion Criteria:

* • Surgical liposuction within the last 12 months.

  * Untreated hypo- or hyperthyroidism.
  * Uncontrolled liver, kidney or cardiovascular disease or diabetes.
  * Implanted pacemaker or metal implant.
  * History of thrombophlebitis, any hematological disease.
  * No past or present neurological and musculoskeletal disorders that will have affected health condition.
  * No smoking and drinking habits.
  * No psychological problems.

Ages: 48 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 4 months
  Outcome measures, HOMA-IR (Homeostasis Model Assessment) will be used to assess insulin resistance. HOMA-IR is a model of interactions between glucose and insulin dynamics that is then used to predict fasting steady-state glucose and insulin concentrations for a wide range of possible combinations of insulin resistance and β-cell function.

SECONDARY OUTCOMES:
ultrasound | 4 months
  Abdominal fat thickness will be assessed by ultrasound (Aplio 500-model TUS-A500, fundamentals (2B77-004EN*M)
BMI by kg/m2 | 4 months
  weight and height will be combined to report BMI in kg/m^2
waist circumferences by tape | 4 months
The surface under the cumulative ranking curve (SUCRA) | 4 months
  The surface under the cumulative ranking curve (SUCRA) was used to rank and compare the effects of different types of exercise. SUCRA values range from 0 to 100, where 100 indicates the best treatment with no uncertainty and 0 indicates the worst treatment with no uncertainty. Thus, higher SUCRA values indicated the better effects of an exercise intervention prior to and after four-month treatment duration for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Mohammed, Principal Investigator — out patient clinic ,faculty of physical therapy ,Cairo university ,Cairo,Egypt
Locations (1):
- Shymaa Mohammed, Cairo, Egypt